CLINICAL TRIAL: NCT00267085
Title: A Pilot Phase II Trial of a Synthetic Tumor-Specific Breakpoint Peptide Vaccine in Patients With Chronic Myeloid Leukemia (CML) and Minimal Residual Disease
Brief Title: Synthetic Vaccine in Patients With Chronic Myeloid Leukemia and Minimal Residual Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BreakThrough Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0392; NCT00392600 (obsolete NCT alias)
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Myeloid Leukemia; Minimal Residual Disease
Keywords: Chronic Myeloid Leukemia; Minimal Residual Disease; Peptide Vaccine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasm, Residual | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CML Vaccine (Experimental): Imatinib mesylate subcutaneously every 2 weeks x 4 weeks, then every three weeks x 1 week, then monthly for 10 months
  Interventions: Biological: Synthetic Tumor-Specific Breakpoint Peptide Vaccine

INTERVENTIONS:
Biological: Synthetic Tumor-Specific Breakpoint Peptide Vaccine — CML vaccine, Imatinib mesylate, subcutaneously every 2 weeks x 4 weeks, then every three weeks x 1 week, then monthly for 10 months
  Other Names: Imatinib mesylate

SUMMARY:
The goal of this clinical research study is to learn if giving 1 of 2 CML (Chronic Myeloid Leukemia) vaccines (CML-VAX B2 or CML-VAX B3) together with imatinib mesylate can decrease or eliminate all evidence of disease in patients who have CML that is in remission after treatment with imatinib mesylate, but who still have small amounts of detectable disease.

DETAILED DESCRIPTION:
Patients who are eligible to take part in this study have already responded well to treatment with imatinib mesylate. Your disease is in what is called a complete cytogenetic remission (i.e., The Philadelphia chromosome is no longer detectable.). However, there is still a small amount of disease that can be detected using the most sensitive techniques available. CML-VAX B2 and CML-VAX B3 are experimental vaccines made from the proteins that cause leukemia cells in CML to behave abnormally. Imatinib mesylate is the standard therapy for CML and blocks the function of this protein.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam and medical history. Blood (about 2 tablespoons) will be collected for routine tests. You will also have a bone marrow aspiration and a chromosome analysis of the number of chromosomes in the bone marrow. To collect a bone marrow aspiration, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

You will also have some additional blood work (about 1 tablespoon) to test the levels of leukemia in your blood. If you agree to participate in this study, this test will be repeated 2 more times, about 2 weeks apart, before you can start vaccination. This is done to get a good measure of the amount of disease you may have.

There are 2 different vaccines that can be used in this study, CML-VAX B2 and CML-VAX B3. If you are found to be eligible to take part in this study, you will only receive one of them. Which one you receive depends on the type of protein your leukemia makes, as these vaccines are specific to each of the 2 most common proteins that may be produced by CML cells.

All participants in this study will receive 1 of the 2 vaccines as well as imatinib mesylate. Imatinib mesylate will continue to be given to you at the dose that you are taking now. The vaccines will be mixed with a substance called montanide. This is a standard procedure with vaccines and is done to try to make it more likely that you will have a good immune response to the vaccines in general.

When the appropriate vaccine is selected for your use, you will receive an injection of the vaccine once every 2 weeks for the first 8 weeks, once 3 weeks later, and then once every month for a total of 15 vaccines in 12 months. You will receive the vaccine at M. D. Anderson. The vaccine will be injected in the arms or the thighs. Two days before each vaccination and again the day of each vaccination, you will receive an injection of a growth hormone called GM-CSF (Leukine). The purpose of this injection is to boost your immune system, in response to the vaccine, to specifically kill your leukemia. This injection is given through a small needle and injected under your skin in your arms or your thighs. You can be taught how to do this for yourself, but you may choose to have it given to you by a member of the study staff.

Every time that you come in for an injection of the vaccine, you will also have a physical exam and have routine blood work done (about 2 tablespoons). Every 3 months while receiving the vaccine you will also have blood drawn (about 1 tablespoon) to test the level of leukemia and to see if you are responding to the vaccine.

You will be taken off study if intolerable side effects occur or your disease comes out of remission. About 2 weeks after the last injection of vaccine, you will have blood drawn (about 1 tablespoon) to test the level of leukemia and to see if you are responding.

This is an investigational study. CML-VAX B2 and CML-VAX B3 are not FDA approved. The vaccine and montanide will be free. Because you are receiving imatinib mesylate as part of your standard of care, you and/or your insurance company or third-party payer will be responsible for the costs of it. If GM-CSF is not covered by your insurance or other third-party payer, it will be provided free of charge. A maximum of 60 patients will take part in this study. A maximum of 20 will be enrolled at M. D. Anderson.

Optional Procedures: If you agree, additional blood tests (about 3 tablespoons each) will be done at about 30 days before the first vaccine, after 6 months and 9 months from the start of vaccination, and (about 10 tablespoons each) on the day of the first vaccine and after 3 months and 2 weeks after the last vaccine to measure the response of your immune system to the vaccine.

If you agree, a skin test will be done where a small amount of the proteins will be injected under your skin for another measure of response of your immune system. If a small nodule develops in the area where you receive this injection, it may represent an immune response. This will be measured by your doctor or your nurse.

You do not have to agree to take part in the optional procedures in order to receive treatment on this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Ph chromosome positive or BCR-ABL-positive CML (as determined by cytogenetics, FISH, or RT-PCR).
2. Patients must have reached their 18th birthday.
3. Patients must have received imatinib therapy for at least 12 months and must not have had changes in their dose of imatinib in the last 6 months. Patients must not have had a continuous interruption of imatinib therapy of greater than 14 days or for a total of 6 weeks in the 6 months prior to enrollment.
4. Patients must be in complete cytogenetic remission confirmed by two marrows, the second being at least one month after the first.
5. Patients must have detectable BCR-ABL transcript levels that are not more than 0.5-log lower than the lowest value obtained in the last 6 months, with at least two values obtained during this period.
6. Karnofsky performance status should be > 70.
7. Adequate organ function defined as: bilirubin <2x upper limit of normal (ULN), creatinine <1.5x ULN, and ALT and AST <2.5x ULN.
8. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
9. Women of childbearing potential (i.e., not post-menopausal 24 months or not surgically sterile) must agree to use effective methods of contraception.

Exclusion Criteria:

1. Patients with a history of accelerated or blast crisis. Accelerated phase is defined as 15 to 30% blasts or >30% blasts plus promyelocytes in the peripheral blood or marrow, >20% basophils, or platelets <100 x 10^9/L, unrelated to therapy. Cytogenetic abnormalities in addition to the Ph chromosome are not considered a defining feature of accelerated phase.
2. Patients with autoimmune disorders or known immune deficiency.
3. Patients receiving immunosuppressive therapy, corticosteroids, chemotherapy, or therapy for CML other than imatinib.
4. Patients receiving any other investigational agents.
5. Patients who are pregnant or breast-feeding.
6. Patients with clinically significant heart disease (New York Heart Association Class III or IV) or other serious intercurrent illnesses, active uncontrolled infections requiring antibiotics or active bleeding.
7. Patients who have undergone major surgery within 28 days before registration, or who have not fully recovered from any other prior major surgery.
8. Patients who have undergone stem cell transplantation.
9. Patients who have received radiation therapy within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 12/2/05 to 7/1/08. All participants registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Eleven participants were registered, one was excluded from study enrollment and did not receive the Chronic Myeloid Leukemia (CML) Vaccine.
Groups:
- CML Vaccine: Imatinib mesylate subcutaneously every 2 weeks x 4 weeks, then every three weeks x 1 week, followed by monthly for 10 months
Period: Overall Study
Arm/Group | CML Vaccine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CML Vaccine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Median (Full Range); unit: years] | 45 [28 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response: One Log Decrease in BCR-ABL
Description: Molecular response defined as reduction by one log of the circulating peripheral blood for reverse transcription polymerase chain reaction (RT-PCR) transcripts of BCR-ABL (tumor-specific oncogenic fusion protein) after two consecutive measurements. RT-PCR performed at 3 month intervals. Response categorized as either 'No Decrease' or 'Decrease' if one log reduction in BCR-ABL detected.
Time Frame: 12 months
Population: All 10 participants on study received treatment and were included in analysis.
Measure: Number; unit: Participants
Arm/Group | CML Vaccine
Number analyzed (Participants) | 10
Participants
  Decrease | 3
  No Decrease | 7

ADVERSE EVENTS:
Time Frame: 2 years 3 months
Arm/Group | CML Vaccine
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CML Vaccine (N=10)
Neck Pain (General disorders) | 1 (1) — Unrelated to study drug.
Back Pain (General disorders) | 1 (1) — Unrelated to study drug.
Nausea (Gastrointestinal disorders) | 1 (1) — Unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CML Vaccine (N=10)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/skin (other) (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 5 (9)
Fever without neutropenia (General disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 10 (31)
Nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (joint) (General disorders) | 2 (2)
Pain (muscle) (General disorders) | 3 (4)
Pain (NOS) (General disorders) | 1 (1)
Pain (Other) (General disorders) | 2 (2)
Pruitis (Skin and subcutaneous tissue disorders) | 5 (8)
rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (3)
Sweating (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No